CLINICAL TRIAL: NCT06932289
Title: Integrating Metabolic and Vascular Sensors to Monitor Cardiometabolic Disorders After Nutrition Interventions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1832799-1
Record Dates: First submitted 2025-01-21; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: NAFLD; metabolic responses; mixed meal challenge
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Diet 1 (one of the three kinds of diets) (Active Comparator): participants will be randomized to diet 1 for 2 weeks. A continuous glucose monitor (CGM) will be placed and the integrated sweat sensor and vascular sensor will be administered.
  Interventions: Dietary Supplement: Mediterranean diet (MED), high-fat/low carb diet (HF/LC), and low-fat diet (LF); Device: The integrated sweat sensor and vascular sensor (wearable); Device: continuous glucose monitor (CGM)
- Diet 2 (one of the two remaining kinds of diets, excluding Diet 1) (Active Comparator): participants will be randomized to diet 2 for 2 weeks. A continuous glucose monitor (CGM) will be placed and the integrated sweat sensor and vascular sensor will be administered.
  Interventions: Dietary Supplement: Mediterranean diet (MED), high-fat/low carb diet (HF/LC), and low-fat diet (LF); Device: The integrated sweat sensor and vascular sensor (wearable); Device: continuous glucose monitor (CGM)
- Diet 3 (the final remaining diet) (Active Comparator): participants will be randomized to diet 3 for 2 weeks. A continuous glucose monitor (CGM) will be placed and the integrated sweat sensor and vascular sensor will be administered.
  Interventions: Dietary Supplement: Mediterranean diet (MED), high-fat/low carb diet (HF/LC), and low-fat diet (LF); Device: The integrated sweat sensor and vascular sensor (wearable); Device: continuous glucose monitor (CGM)
- Habitual diet as a baseline (Experimental): All participants will consume their habitual diet for 2 weeks to establish baseline. A continuous glucose monitor (CGM) will be placed and the integrated sweat sensor and vascular sensor will be administered.
  Interventions: Device: The integrated sweat sensor and vascular sensor (wearable); Device: continuous glucose monitor (CGM)

INTERVENTIONS:
Dietary Supplement: Mediterranean diet (MED), high-fat/low carb diet (HF/LC), and low-fat diet (LF) — Participants will be randomized to either Mediterranean diet (MED), high-fat/low carb diet (HF/LC), or low-fat diet (LF).
  Arms: Diet 1 (one of the three kinds of diets); Diet 2 (one of the two remaining kinds of diets, excluding Diet 1); Diet 3 (the final remaining diet)
Device: The integrated sweat sensor and vascular sensor (wearable) — The integrated sweat sensor and vascular sensor will be worn of each diet period.
Device: continuous glucose monitor (CGM) — A continuous glucose monitor (CGM) will be placed on the patients during each diet period.

SUMMARY:
It is a 12-week study. The participants will follow three different diets, and during each diet period, and the participants will wear our device, and blood samples will be collected.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, controlled crossover intervention study. The investigators will enroll 54 participants, aged >18 years, BMI >25 kg/m2 with metabolic syndrome. During the first phase, all participants will consume their habitual diet for 2 weeks to establish baseline. Then participants will be randomized to either a Mediterranean diet (MED), high-fat/low carb diet (HF/LC), or low-fat diet (LF) for 14 days with 2 weeks washout between the different diets. The wearable system will monitor basal levels and the changes for glucose, cholesterol, TG, and NO through sweat analysis and HR, HRV, and PWV for carotid arterial stiffness during each diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* United States Veterans
* Male or female, age 18-55 years at the time of signing informed consent.
* at least 2 of the following: waist circumference > 40" for men and 35" for women, FBS >100 mg/dl, triglycerides > 150 but < 500 mg/dL, HDL < 40 mg/dL, Pre- hypertension or hypertension (BP>120/80 mmHg but <150/90 mmHg)

Exclusion Criteria:

* History of diabetes require medications
* History of alcohol intake ≥ 20g/day
* History of cirrhosis
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of <30 mL/min/1.73 m2
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* Any unstable medical conditions or terminal diagnosis.
* Any participant who is unwilling to sign an informed consent form will not be admitted into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of glucose | From enrollment to the end of measurement at 12 weeks
  The concentration of glucose (mg/dL) will be measured during each visit, across the different diets, to evaluate changes in metabolism
Concentration of cholesterol | From enrollment to the end of measurement at 12 weeks
  The concentration of cholesterol (mg/dL) will be measured during each visit, across the different diets, to evaluate changes in metabolism.
Concentration of triacylglycerol (TG) | From enrollment to the end of measurement at 12 weeks]
  The concentration of triacylglycerol (TG) (mg/dL) will be measured during each visit, across the different diets, to evaluate changes in metabolism.
Concentration of Nitric oxide (NO) | From enrollment to the end of measurement at 12 weeks
  The concentration of Nitric oxide (NO) (ppm) will be measured during each visit, across the different diets, to evaluate changes in metabolism.
Measurement of heart rate (HR) | From enrollment to the end of measurement at 12 weeks
  The heart rate (HR) (bpm) will be measured during each visit, across the different diets, to evaluate changes in vessel stiffness indirectly.
Measurement of heart rate variability (HRV) | From enrollment to the end of measurement at 12 weeks
  The heart rate variability (HRV) (ms) will be measured during each visit, across the different diets, to evaluate changes in vessel stiffness indirectly.
Measurement of pulse wave velocity (PWV) | From enrollment to the end of measurement at 12 weeks
  The pulse wave velocity (PWV) (m/s) will be measured during each visit, across the different diets, to evaluate changes in vessel stiffness.
Body weight | From enrollment to the end of measurement at 12 weeks
  The body weight (BW) (kg) will be measured during each visit, across the different diets, to evaluate changes of BMI.
Height | From enrollment to the end of measurement at 12 weeks
  The height (m) will be measured during each visit, across the different diets, to evaluate changes in BMI.

SECONDARY OUTCOMES:
BMI | From enrollment to the end of measurement at 12 weeks
  The Body mass index (BMI) (kg/m2) will be measured during each visit, across the different diets, to evaluate changes of body fat.

CONTACTS AND LOCATIONS:
Overall Officials: Tzung Hsiai, M.D., Ph.D., Principal Investigator — VAGLAHS and UCLA
Locations (1):
- Va Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The results of a research study may be published in the medical literature or presented at scientific medical or educational meetings, but the Veteran participant's name or identity will not be revealed, and their records will remain confidential unless disclosure of your identity is required by law.